CLINICAL TRIAL: NCT06957223
Title: Efficacy of Dextromethorphan-Bupropion Versus SSRIs in the Treatment of Major Depressive Disorder: A Randomized Controlled Trial
Brief Title: Efficacy of Dextromethorphan-Bupropion Versus SSRIs in the Treatment of Major Depressive Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asad Ullah Jan (Other Government)
Collaborators: CMH Nowshera (Unknown)
Responsible Party: Sponsor-Investigator, Asad Ullah Jan, Head Department of Psychiatry, Combined Military Hospital Nowshera
Organization: Combined Military Hospital Nowshera (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMHNSR-REF-16
Record Dates: First submitted 2025-04-26; First posted 2025-05-04 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dextromethorphan-Bupropion Group (Experimental): Participants will receive a fixed-dose combination of dextromethorphan-bupropion, dosed according to approved guidelines for major depressive disorder, administered orally for 6 weeks.
  Interventions: Drug: Dextromethorphan-Bupropion
- SSRI Group (Active Comparator): Participants will receive an SSRI at standard therapeutic doses, administered orally for 6 weeks.
  Interventions: Drug: SSRIs

INTERVENTIONS:
Drug: Dextromethorphan-Bupropion — Participants will receive a fixed-dose combination of dextromethorphan-bupropion, dosed according to approved guidelines for major depressive disorder, administered orally for 6 weeks.
  Arms: Dextromethorphan-Bupropion Group
Drug: SSRIs — Participants will receive an SSRI at standard therapeutic doses, administered orally for 6 weeks.
  Arms: SSRI Group

SUMMARY:
The study aims to compare the antidepressant effects of a dextromethorphan-bupropion combination versus standard SSRI therapy in adult patients with major depressive disorder. Participants will be randomized into two groups: one receiving dextromethorphan-bupropion and the other receiving an SSRI (e.g., sertraline or escitalopram). Treatment will last for 6 weeks, with assessments at baseline and study completion. The primary outcome will be the remission rate measured by a validated depression rating scale. Secondary outcomes include change in depressive symptoms severity and safety/tolerability measures.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with major depressive disorder (MDD) per DSM-5 criteria.

Baseline depression score indicating moderate to severe depression

Ability to provide informed consent

Willing to comply with study requirements

Exclusion Criteria:

History of bipolar disorder, schizophrenia, or other psychotic disorders

Current substance use disorder (within past 6 months)

Active suicidal ideation requiring urgent intervention

Pregnancy or breastfeeding

Known hypersensitivity to study medications

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2025-05-06 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Depression Severity (measured by HAMD-17) | 6 weeks
  Change from baseline in depressive symptom scores, measured using the Hamilton Depression Rating Scale, 17-item version (HAMD-17; score range 0-52, with higher scores indicating worse depression severity).

SECONDARY OUTCOMES:
Remission Rate | 6 weeks
  Proportion of participants achieving remission, defined as a depression rating scale score below the clinical threshold.

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Combined Military Hospital, Nowshera, KPK
  - Department of Psychiatry, Combined Military Hospital Nowshera, Nowshera, KPK

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to confidentiality concerns and lack of infrastructure for data sharing.